CLINICAL TRIAL: NCT02760147
Title: Evaluation of Beacon Care System Advice in Pressure Support: Does the System Maintain Patients Within Appropriate Levels of Support?
Brief Title: BEACON Care ® System Assisting Ventilation in Pressure Support Ventilation (PSV) Patient
Acronym: BEACON3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Assistant Professor - Researcher, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20150604
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Artificial Respiration
Keywords: Pressure Support Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pressure Support Over Support (Other): Pressure Support Level upward by 50%, 2 hours
  Interventions: Device: Pressure Support Over Support; Device: Pressure Support Under Support
- Pressure Support Under Support (Other): Pressure Support Level downward by 50%, 2 hours
  Interventions: Device: Pressure Support Over Support; Device: Pressure Support Under Support
- PEEP Over Level (Other): PEEP Level upward by 50%, 2 hours
  Interventions: Device: PEEP Over Level; Device: PEEP Under Level
- PEEP Under Level (Other): PEEP Level downward by 50%, 2 hours
  Interventions: Device: PEEP Over Level; Device: PEEP Under Level

INTERVENTIONS:
Device: Pressure Support Over Support — Pressure Support Level upward by 50%, 2 hours
  Arms: Pressure Support Over Support; Pressure Support Under Support
Device: Pressure Support Under Support — Pressure Support Level downward by 50%, 2 hours
  Arms: Pressure Support Over Support; Pressure Support Under Support
Device: PEEP Over Level — PEEP Level upward by 50%, 2 hours
  Arms: PEEP Over Level; PEEP Under Level
Device: PEEP Under Level — PEEP Level downward by 50%, 2 hours
  Arms: PEEP Over Level; PEEP Under Level

SUMMARY:
The aim of this study is to evaluate the ventilator settings advice given by the BEACON care system in fitting with best level of support in patient under mechanical ventilation in Pressure Support mode.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether pressure support settings suggested by the B3 system and pressure support as well as Positive End Expiratory Pressure (PEEP) settings suggested by the B5 system, i.e. balancing under and over support based upon physiological models and simple clinical measures, are consistent with keeping patients within appropriate levels of support as assessed by the ratio between airwaiy pressure generated by the respiratory muscles (Pmus) and the maximum inspiratory pressure (MIP) (Pmus/MIP), the ratio between the inspiratory time (TI) and total respiratory time (TTOT) (TI/TTOT) and the Tension-Time index (TTi), these being obtained using less frequently used esophageal catheter measurements.

ELIGIBILITY:
Inclusion Criteria:

* Under mechanical ventilation in Pressure Support mode

Exclusion Criteria:

* Neuromuscular impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reduction of respiratory fatigue of patient under mechanical ventilation | Average of 1 hour
  Esophageal catheter will be positioned and pressure generated by the respiratory muscles will be measured to detect respiratory muscles' fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Rees, Medical, Study Director — Aalborg University; Dan Stieper Karbing, Engenieer, Principal Investigator — Aalborg University; Savino Spadaro, Medicine, Principal Investigator — Ferrara University; Carlo Alberto Volta, Medicine, Study Director — Ferrara University
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No